CLINICAL TRIAL: NCT02516215
Title: Population Research of Sublingual Microcirculation Data of Patients With Systemic Diseases
Brief Title: Sublingual Microcirculation Data of Patients With Systemic Diseases
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201505008RINA
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Sublingual Microcirculation Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (8):
- 1_Hypertension: Patients with diagnosed hypertension, without other systemic diseases
  Interventions: Other: No intervention
- 2_Diabetes mellitus: Patients with diagnosed diabetes mellitus, without other systemic diseases
  Interventions: Other: No intervention
- 3_Hypertension and diabetes mellitus: Patients with both diagnosed hypertension and diabetes mellitus
  Interventions: Other: No intervention
- 4_end stage renal disease with hemodialysis: Patients with end stage renal disease with hemodialysis
  Interventions: Other: No intervention
- 5_Peripheral arterial occlusive disease: Patients with disgnosed peripheral arterial occlusive disease
  Interventions: Other: No intervention
- 6_Coronary artery disease: Patients with diagnosed coronary artery disease
  Interventions: Other: No intervention
- 7_liver cirrhosis: Patients with diagnosed liver cirrhosis
  Interventions: Other: No intervention
- 8_Anemia: Patients with diagnosed anemia
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
This is an observational clinical study, patients with systemic diseases will be enrolled according to the inclusion and exclusion criteria. 360 patients will received the examination of sublingual microcirculation by using sidestream dark filed video microscope. The microcirculation data includes total small vessel density, perfused small vessel density, microvascular flow index, and heterogeneity index. The patients will be divided into right groups according to their systemic diseases as follows: group 1 hypertension (60 patients), group 2 diabetes mellitus (60), group 3 hypertension and diabetes mellitus (60), group 4 end stage renal disease with hemodialysis (60), group 5 peripheral arterial occlusive disease (30), group 6 coronary artery disease (30), group 7 liver cirrhosis (30), and group 8 anemia (30).

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 20 to 79 years old
* BMI ranged from 18.5 to 27 kg/m2
* Presence of one of the condition

  1. Diagnosed hypertenison > 6 months, without other systemic diseases
  2. Diagnosed diabetes mellitus > 6 monthes, without other systemic diseases
  3. Diagnosed with both hypertension and diabetes mellitus > 6 months, without other systemic diseases
  4. Diagnosed with end stage renal disease and recevied renal replacement therapy > 6 months
  5. Diagnosed with peripheral arterial occlusive diseases > 6 months
  6. Diagnosed with coronary artery disease > 6 months
  7. Diagnosed with liver cirrhosis > 6 months
  8. Diagnosed with anemia > 6 months, hemoglobin level < 10 g/dL

Exclusion Criteria:

* Diagnosed with sepsis, major tauma, or admission to ICU within one month
* Body temperature higher than 37.5 ℃ or lower than 35.5 ℃
* Any on of the following condition

  1. Asthma
  2. Chronic obstructive pulmonary disease
  3. Endocrine diseases
  4. Hematological disorders
  5. Uncured cancer
  6. Chronic uncured infection
  7. Other major disease with limited daily activity
* Non-native speakers

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diagnosed hypertension, diabetes mellitus, both hypertension and diabetes mellitus, end stage renal disease with hemodialysis, peripheral arterial occlusive disease, coronary artery disease, liver cirrhosis, or anemia.
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Total small vessel density of sublingual small vessels | Once at enrollment
  Total small vessel density will be measured by Microscan and analyzed by AVA 3.0 software

SECONDARY OUTCOMES:
Perfused small vessel density of sublingual small vessels | Once at enrollment
  Perfused small vessel density will be measured by Microscan and analyzed by AVA 3.0 software

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chang Yeh, M.D., Ph.D., Principal Investigator — National Taiwan University Hospital, Department of Anesthesiology
Locations (1):
- National Taiwan University Hospital, anesthesiology department, Taipei, Taiwan